CLINICAL TRIAL: NCT02788513
Title: A Multi-centre, Double-blind, Parallel-group, Randomised Controlled Study to Investigate Efficacy and Safety of Orally Administered BI 425809 During a 12-week Treatment Period Compared to Placebo in Patients With Cognitive Impairment Due to Alzheimer's Disease.
Brief Title: BI 425809 in Patients With Cognitive Impairment Due to Alzheimer's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1346.23; 2015-005438-24 (EudraCT Number)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BI 425809 dose 1 (Experimental)
  Interventions: Drug: BI 425809 dose 1; Drug: Placebo
- BI 425809 dose 2 (Experimental)
  Interventions: Drug: BI 425809 dose 2; Drug: Placebo
- BI 425809 dose 3 (Experimental)
  Interventions: Drug: BI 425809 dose 3; Drug: Placebo
- BI 425809 dose 4 (Experimental)
  Interventions: Drug: BI 425809 dose 4; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 425809 dose 1
  Arms: BI 425809 dose 1
Drug: BI 425809 dose 2
  Arms: BI 425809 dose 2
Drug: BI 425809 dose 3
  Arms: BI 425809 dose 3
Drug: BI 425809 dose 4
  Arms: BI 425809 dose 4
Drug: Placebo

SUMMARY:
The study is designed to compare the effects of BI 425809 compared to placebo in patients with cognitive impairment due to Alzheimer's Disease.

ELIGIBILITY:
Inclusion criteria:

* Patients with early signs of dementia of Alzheimer Type
* Male and female patients with an age of at least 55 years
* Concomitant use of acetylcholinesterase inhibitors (AChEIs) is allowed but not required. Patients who are currently taking AChEIs are eligible as long as they have been using a stable dose for at least 3 months prior to screening and no change is foreseen for the duration of the study. This dose must be consistent with the product label in the concerned country. Patients who are not currently taking AChEIs but have taken them in the past are also eligible if AChEIs were stopped at least 3 months prior to screening.
* Patients must have at least 6 years of formal education and fluency in the test language as verbally confirmed by the patient and documented by the study investigator.
* Patients must have a reliable study partner (per investigator judgement, for instance a family member, partner etc., guardian)
* Further inclusion criteria apply

Exclusion criteria:

* Cognitive impairment or dementia with any etiology other than Alzheimer's Dementia (AD)
* Substantial concomitant cerebrovascular disease (defined by a history of a stroke / intracranial haemorrhagia) temporally related to the onset of worsening of cognitive impairment per investigator judgement
* Medical history or diagnosis of any of symptomatic and unstable/uncontrolled conditions per investigator judgement
* Patients receiving prescribed drugs for treatment of dementia of Alzheimer Type (other than Acetylcholine Esterase Inhibitors) at screening or within 3 months prior to screening
* Previous participation in investigational drug studies of dementia of Alzheimer's Type within three months prior to screening. Patients having received any active treatment in studies targeting disease modification of AD are excluded. Previous participation in studies with non-prescription medications, vitamins or other nutritional formulations is allowed.
* Clinically significant uncompensated hearing loss in the judgment of the investigator. Use of hearing aids is allowed.
* Further exclusion criteria apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (93):
- United States (17):
  - Axiom Research LLC, Colton, California
  - Alliance for Wellness, Long Beach, California
  - Anderson Clinical Research, Redlands, California
  - CITrials, Santa Ana, California
  - MD Clinical, Hallandale, Florida
  - Galiz Research, Miami, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Miami Jewish Health System, Miami, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Bioclinica Research, The Villages, Florida
  - Neuro Trials Research Incorporated, Atlanta, Georgia
  - Millennium Psychiatric Associates LLC, St Louis, Missouri
  - ANI Neurology, PLLC, dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Northeastern Pennsylvania Memory and Alzheimer Center, Plains, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - The Memory Clinic, Bennington, Vermont
- Austria (4):
  - LKH-Univ. Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - SALK Christian-Doppler-Klinik,Paracel.Med.Privatuni.f.Neurol, Salzburg
  - Private Practice for Psychiatry and Neurology, Vienna
- Canada (6):
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - True North Clinical Research Halifax, Inc., Halifax, Nova Scotia
  - True North Clinical Research Kentville, Inc., Kentville, Nova Scotia
  - Bluewater Clinical Research, Sarnia, Ontario
  - Clinique Neuro-Outaouais, Gatineau, Quebec
  - Diex Recherche, Sherbrooke, Quebec
- Finland (5):
  - Orton, Helsinki
  - University of Eastern Finland, Brain Research Unit, Kuopio
  - Terveystalo Lahti, Lahti
  - OYS, Neurologian tutkimusyksikkö, Oulu
  - CRST - Clinical Research Services Turku, Turku
- France (9):
  - HOP Pellegrin, Bordeaux
  - HOP Pierre Wertheimer, Bron
  - HOP Roger Salengro, Lille
  - HOP Gui de Chauliac, Montpellier
  - HOP Nord Laënnec, Nantes
  - HOP La Pitié Salpêtrière, Paris
  - CHU La Grave-Casselardit - Cité de la Santé, Toulouse
  - HOP Brabois, Vandœuvre-lès-Nancy
  - HOP des Charpennes, Villeurbanne
- Germany (8):
  - Zentrum für klinische Forschung Dr. med. Irma Schöll & Kollegen, Bad Homburg
  - Praxis Dr. med. Volker Schumann, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Praxis Dr. Oehlwein, Gera
  - Pharmakologisches Studienzentrum Chemnitz, Mittweida
  - Institut für Psychogerontologie, Nuremberg
  - Neuropraxis München Süd, Unterhaching, Unterhaching
- Greece (5):
  - Naval Hospital of Athens, Athens
  - Eginition Hospital, Athens
  - University General Hospital Attikon, Athens
  - Athens Medical Center, Athens
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Hungary (3):
  - Semmelweis University, Budapest
  - CRU Ltd, Neurology Dept., Miskolc, Miskolc
  - University of Szeged, Szeged
- Italy (4):
  - IRCCS Fondazione Ospedale Maggiore, Milan
  - A.O. San Gerardo di Monza, Monza (MB)
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Japan (12):
  - Fujita Health University Hospital, Aichi, Toyoake
  - Inage Neurology and Memory Clinic, Chiba, Chiba
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Kawashima Neurology Clinic, Kanagawa, Fujisawa
  - Ishikawa Clinic, Kyoto, Kyoto
  - Nara Medical University Hospital, Nara, Kashihara
  - Katayama Medical Clinic, Okayama, Kurashiki
  - National Hospital Organization Hizen Psychiatric Center, Saga, Kanzaki-gun
  - National Center Neurology and Psychiatry, Tokyo, Kodaira
  - Nozomi Memory Clinic, Tokyo, Mitaka
  - Showa University East Hospital, Tokyo, Shinagawa
- Norway (2):
  - Oslo Universitetssykehus HF, Hukommelsesklinikken, Oslo
  - St. Olavs Hospital, Universitetssykehuset i Trondheim, Trondheim
- Poland (5):
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Non-Public Outpat. Clinic "Dom Sue Ryder", PALLMED Sp. z o.o, Bydgoszcz
  - Non-Public Outpatient Clinic Neuro-Kard Ilkowski & Partners, Poznan
  - EUROMEDIS Sp. z o.o., Szczecin, Szczecin
  - Clin.Research Centre Clinsante SC Ewa Galczak-Nowak,Torun, Torun
- Spain (6):
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu de Manresa, Manresa
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Viamed Montecanal, Zaragoza
- United Kingdom (7):
  - Royal Cornhill Hospital, Aberdeen
  - Fulbourn Hospital, Cambridge
  - Ninewells Hospital & Medical School, Dundee
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Warneford Hospital, Oxford
  - Sheffield Memory Service, Sheffield

REFERENCES:
- [Derived] Wunderlich G, Blahova Z, Garcia M, Jessen F. Efficacy and safety of the novel GlyT1 inhibitor BI 425809 in Alzheimer's dementia: a randomized controlled trial. Alzheimers Res Ther. 2023 Jan 28;15(1):24. doi: 10.1186/s13195-023-01163-3. PMID 36709275
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multi-centre, double-blind, parallel-group, randomised controlled study to investigate efficacy and safety of orally administered BI 425809 during a 12-week treatment period compared to placebo in patients with cognitive impairment due to Alzheimer's Disease.
Pre-assignment Details: Subjects were screened prior to participation and attended a specialist site which ensured that they strictly met all inclusion/exclusion criteria. Subjects were not to be allocated to a treatment group if any of the criteria were violated.
  One subject was randomized by error via Interactive Response Technology (IRT) but never took a drug.
Groups:
- 2 mg BI 425809: Participants in dose group 1 were orally administered 2 tablets of 1 milligrams (mg) of BI 425809 (Total: 2 mg) together with 1 tablet of 25 mg placebo match once daily (qd) during 12 weeks. The tablets were to be taken with water in the morning at approximately the same time every day with or without food.
- 5 mg BI 425809: Participants in dose group 2 were orally administered 1 tablet of 5 mg of BI 425809 together with 1 tablet of 1 mg / 5 mg and 1 tablet of 25 mg placebo match once daily (qd) during 12 weeks. The tablets were to be taken with water in the morning at approximately the same time every day with or without food.
- 10 mg BI 425809: Participants in dose group 3 were orally administered 2 tablets of 5 mg of BI 425809 (Total: 10 mg) together with 1 tablet of 25 mg placebo match once daily (qd) during 12 weeks. The tablets were to be taken with water in the morning at approximately the same time every day with or without food.
- 25 mg BI 425809: Participants in dose group 4 were orally administered 1 tablet of 25 mg of BI 425809 together with 2 tablets of 1 mg / 5 mg of placebo match once daily (qd) during 12 weeks. The tablets were to be taken with water in the morning at approximately the same time every day with or without food.
- Placebo Group: Participants in the placebo group were orally administered 2 tablets of 1 mg / 5 mg and 1 tablet of 25 mg of placebo match once daily (qd) during 12 weeks. The tablets were to be taken with water in the morning at approximately the same time every day with or without food.
Period: Overall Study
Arm/Group | 2 mg BI 425809 | 5 mg BI 425809 | 10 mg BI 425809 | 25 mg BI 425809 | Placebo Group
Started | 123 | 122 | 122 | 123 | 120
Completed | 114 | 114 | 114 | 117 | 115
Not Completed | 9 | 8 | 8 | 6 | 5
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 5 | 8 | 4 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0
Not completed — Subject decided to stop taking treatment | 0 | 0 | 1 | 0 | 0
Not completed — Decision by the study team | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): the TS included all patients treated with at least one dose of trial medication. Patients in the treated set were analysed based on the actual treatment received at the randomisation. The TS was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 mg BI 425809 | 5 mg BI 425809 | 10 mg BI 425809 | 25 mg BI 425809 | Placebo Group | Total
Number analyzed (Participants) | 123 | 122 | 122 | 123 | 120 | 610
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (7.5) | 72.5 (8.2) | 74.4 (6.9) | 72.9 (7.7) | 72.4 (7.9) | 72.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 62 | 66 | 64 | 64 | 324
  Male | 55 | 60 | 56 | 59 | 56 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 22 | 11 | 16 | 20 | 86
  Not Hispanic or Latino | 101 | 98 | 106 | 103 | 94 | 502
  Unknown or Not Reported | 5 | 2 | 5 | 4 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 11 | 10 | 12 | 14 | 11 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 1 | 1 | 2 | 6
  Black or African American | 10 | 5 | 4 | 3 | 8 | 30
  White | 97 | 103 | 100 | 102 | 93 | 495
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 5 | 3 | 6 | 21
ADASCOG baseline cognitive assessment data [Mean (Standard Deviation); unit: score on a scale] — The Alzheimer's Disease Assessment Scale-Cognitive subscale 11 item (ADAS-Cog11) is an 11-item cognitive subscale that objectively measures memory, language, orientation and praxis with a total score range of 0 to 70, with lower scores indicating less severe impairment. A negative change indicates an improvement from baseline. Population: Treated set (TS): the TS included all patients treated with at least one dose of trial medication. Patients in the treated set were analysed based on the actual treatment received at the randomisation. The TS was used for safety analyses. One placebo subject was without baseline measures due to study was put on hold.
  score on a scale
    number analyzed (Participants) | 123 | 122 | 122 | 123 | 119 | 609
    (all) | 18.8 (7.9) | 18.8 (7.4) | 19.6 (7.8) | 19.6 (7.3) | 18.2 (8.0) | 19.0 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 Item (ADAS-Cog11) Total Score After 12 Weeks of Treatment
Description: The ADAS-Cog11 is an 11-item cognitive subscale that objectively measures memory, language, orientation and praxis with a total score range of 0 to 70, with lower scores indicating less severe impairment. A negative change indicates an improvement from baseline.
  Multiple comparison procedures and modelling (MCPmod) in combination with mixed model repeated measures (MMRM) is used for primary analysis of the primary endpoint.
  MMRM included fixed, categorical covariates of treatment, visit, baseline Mini Mental State Examination MMSE (>=20, <20) and treatment-by-visit interaction, as well as the continuous fixed covariates of baseline and baseline-by-visit interaction. Patient was considered as random effect. The unstructured covariance structure was used to model the within patient measurements. The same MMRM model used in the primary analysis is used for the secondary analysis of the primary endpoint.
Time Frame: On day 1 (visit 2, baseline) and day 85 (end of trial)
Population: Full analysis set (FAS): all randomised patients who were treated with at least one dose of trial medication and had a baseline and at least one corresponding post-baseline on-treatment efficacy assessment for any efficacy endpoint. FAS was used for efficacy analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2 mg BI 425809 | 5 mg BI 425809 | 10 mg BI 425809 | 25 mg BI 425809 | Placebo Group
Number analyzed (Participants) | 121 | 120 | 121 | 119 | 118
score on a scale | 0.026 (4.864) | 0.175 (4.471) | 0.699 (4.313) | -0.174 (4.044) | 0.138 (4.939)
Statistical Analysis 1: Comparison: 2 mg BI 425809 vs 5 mg BI 425809 vs 10 mg BI 425809 vs 25 mg BI 425809 vs Placebo Group; Multiple comparison procedures and modelling (MCPmod) techniques for mixed model repeated measures (MMRM) was used; Test type: Other; p = 0.9931, MCPMod Beta model fit. — An alpha of 0.05 was used for one-sided test. The MCPMod procedure adjusts for multiplicity; Model assumption: 75% of max effect is achieved at 2 mg, 87.5% at 5 mg, 25% at 25 mg, max effect achieved at 10 mg of BI 425809, scalar parameter = 26
Statistical Analysis 2: Comparison: 2 mg BI 425809 vs 5 mg BI 425809 vs 10 mg BI 425809 vs 25 mg BI 425809 vs Placebo Group; Multiple comparison procedures and modelling (MCPmod) techniques for mixed model repeated measures (MMRM) was used; Test type: Other; p = 0.9225, MCPMod Emax model fit. — An alpha of 0.05 was used for one-sided test. The MCPMod procedure adjusts for multiplicity; Model assumption: 20% of the maximum effect is achieved at 2 mg
Statistical Analysis 3: Comparison: 2 mg BI 425809 vs 5 mg BI 425809 vs 10 mg BI 425809 vs 25 mg BI 425809 vs Placebo Group; Multiple comparison procedures and modelling (MCPmod) techniques for mixed model repeated measures (MMRM) was used; Test type: Other; p = 0.9287, MCPMod Sigmoidal Emax model fit. — An alpha of 0.05 was used for one-sided test. The MCPMod procedure adjusts for multiplicity; Model assumption: 25% of max effect achieved at 5 mg and 75% of max effect achieved at 10 mg of BI 425809
Statistical Analysis 4: Comparison: 2 mg BI 425809 vs 5 mg BI 425809 vs 10 mg BI 425809 vs 25 mg BI 425809 vs Placebo Group; Multiple comparison procedures and modelling (MCPmod) techniques for mixed model repeated measures (MMRM) was used; Test type: Other; p = 0.7646, MCPMod linear model fit. — An alpha of 0.05 was used for one-sided test. The MCPMod procedure adjusts for multiplicity; No assumption needed
Statistical Analysis 5: Comparison: 2 mg BI 425809 vs 5 mg BI 425809 vs 10 mg BI 425809 vs 25 mg BI 425809 vs Placebo Group; Multiple comparison procedures and modelling (MCPmod) techniques for mixed model repeated measures (MMRM) was used; Test type: Other; p = 0.9335, MCPMod linear in log model fit. — An alpha of 0.05 was used for one-sided test. The MCPMod procedure adjusts for multiplicity; No assumption needed
Statistical Analysis 6: Comparison: 2 mg BI 425809 vs 5 mg BI 425809 vs 10 mg BI 425809 vs 25 mg BI 425809 vs Placebo Group; Multiple comparison procedures and modelling (MCPmod) techniques for mixed model repeated measures (MMRM) was used; Test type: Other; p = 0.8199, MCPMod logistic model fit. — An alpha of 0.05 was used for one-sided test. The MCPMod procedure adjusts for multiplicity; Model assumption: 10% of max effect achieved at 5 mg and 50% of max effect achieved at 10 mg of BI 425809
Statistical Analysis 7: Comparison: 2 mg BI 425809 vs Placebo Group; Mixed model repeated measures (MMRM); Test type: Other; p = 0.9340, MMRM — p-values are nominal without multiplicity adjustment; MMRM information is described in the description section; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.09 to 1.18], Standard Error of Mean 0.58
Statistical Analysis 8: Comparison: 5 mg BI 425809 vs Placebo Group; Mixed model repeated measures (MMRM); Test type: Other; p = 0.6041, MMRM — p-values are nominal without multiplicity adjustment; MMRM information is described in the description section; Median Difference (Final Values) = 0.30, 95% CI 2-sided [-0.84 to 1.44], Standard Error of Mean 0.58
Statistical Analysis 9: Comparison: 10 mg BI 425809 vs Placebo Group; Mixed model repeated measures (MMRM); Test type: Other; p = 0.1926, MMRM — p-values are nominal without multiplicity adjustment; MMRM information is described in the description section; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-0.38 to 1.90], Standard Error of Mean 0.58
Statistical Analysis 10: Comparison: 25 mg BI 425809 vs Placebo Group; Mixed model repeated measures (MMRM); Test type: Other; p = 0.9739, MMRM — p-values are nominal without multiplicity adjustment; MMRM information is described in the description section; Median Difference (Final Values) = -0.02, 95% CI 2-sided [-1.16 to 1.12], Standard Error of Mean 0.58

2. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS-ADL) Score After 12 Weeks of Treatment
Description: Change from baseline in the ADCS-ADL score after 12 weeks of treatment is presented.
  The ADCS-ADL is a rating scale used to assess basic and instrumental activities of daily living. In the full version of the scale, 23 items are rated by the investigator using information supplied by the caregiver. Each item has a score range varying from 0-3 to 0-5. The sum score could range from 0 to 78, with higher scores indicating less severe impairment. A positive change indicates an improvement from baseline.
  Abbreviation: MMSE = Mini Mental State Examination
Time Frame: On day 1 (visit 2, baseline) and day 85 (end of trial)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2 mg BI 425809 | 5 mg BI 425809 | 10 mg BI 425809 | 25 mg BI 425809 | Placebo Group
Number analyzed (Participants) | 113 | 111 | 110 | 116 | 111
score on a scale | 0.283 (6.805) | 0.577 (5.852) | -1.145 (4.764) | -1.828 (7.034) | 0.261 (4.842)
Statistical Analysis 1: Comparison: 2 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.979, ANCOVA — p-values are nominal without multiplicity adjustment; Analysis of Covariance model included baseline value for the secondary endpoint measure, MMSE stratification (>=20, <20) at baseline and treatment; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-1.48 to 1.52], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: 5 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.521, ANCOVA — p-values are nominal without multiplicity adjustment; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-1.01 to 2.00], Standard Error of Mean 0.77
Statistical Analysis 3: Comparison: 10 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.047, ANCOVA — p-values are nominal without multiplicity adjustment; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-3.04 to -0.02], Standard Error of Mean 0.77
Statistical Analysis 4: Comparison: 25 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.005, ANCOVA — p-values are nominal without multiplicity adjustment; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-3.65 to -0.67], Standard Error of Mean 0.76

3. Secondary Outcome: Clinician's Interview-Based Impression of Change (CIBIC+) Score After 12 Weeks of Treatment
Description: Clinician's Interview-Based Impression of Change (CIBIC+) score is based on semi-structured interview covering domains of function and cognition. It additionally requires the assessment of psychiatric signs and symptoms. The patient and their caregiver are interviewed and questioned by the clinician. Change rate is based on an unanchored 7-point scale (with 0 being not assessed, 1-3 being very much improved to minimally improved, 4 being no change, and 5-7 being minimally worse to very much worse).
  For the ANCOVA model, the baseline value for CIBIC+ is represented by CIBIS which is clinician's interview-based impression of severity score (scores range from 0-7, with 0 being not assessed, 1 being normal, and 7 being most extremely ill) in order to adjust for potential baseline heterogeneity.
  Abbreviation: MMSE = Mini Mental State Examination
Time Frame: On day 1 (visit 2, baseline) and day 85 (end of trial)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2 mg BI 425809 | 5 mg BI 425809 | 10 mg BI 425809 | 25 mg BI 425809 | Placebo Group
Number analyzed (Participants) | 114 | 112 | 110 | 116 | 112
score on a scale | 4.000 (0.941) | 4.080 (0.773) | 4.209 (0.679) | 4.224 (0.781) | 4.080 (0.829)
Statistical Analysis 1: Comparison: 2 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.343, ANCOVA — p-values are nominal without multiplicity adjustment; ANCOVA included MMSE stratification (>=20, <20) at baseline (BL) and treatment, CIBIS is included as BL adjustment term; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.32 to 0.11], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: 5 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.645, ANCOVA — p-values are nominal without multiplicity adjustment; ANCOVA included MMSE stratification (>=20, <20) at baseline (BL) and treatment, CIBIS is included as BL adjustment term; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.26 to 0.16], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: 10 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.448, ANCOVA — p-values are nominal without multiplicity adjustment; ANCOVA included MMSE stratification (>=20, <20) at baseline (BL) and treatment, CIBIS is included as BL adjustment term; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.13 to 0.30], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: 25 mg BI 425809 vs Placebo Group; Analysis of Covariance (ANCOVA); Test type: Other; p = 0.340, ANCOVA — p-values are nominal without multiplicity adjustment; ANCOVA included MMSE stratification (>=20, <20) at baseline (BL) and treatment, CIBIS is included as BL adjustment term; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.11 to 0.32], Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of treatment + 28 days of follow-up, up to 16 weeks.
Description: Treated set (TS): the TS included all patients treated with at least one dose of trial medication. Patients in the treated set were analysed based on the actual treatment received at the randomisation.
Arm/Group | 2 mg BI 425809 | 5 mg BI 425809 | 10 mg BI 425809 | 25 mg BI 425809 | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/122 | 0/122 | 0/123 | 0/120
Serious Adverse Events (participants affected / at risk) | 5/123 | 4/122 | 4/122 | 4/123 | 5/120
Other Adverse Events (participants affected / at risk) | 17/123 | 22/122 | 14/122 | 19/123 | 12/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg BI 425809 (N=123) | 5 mg BI 425809 (N=122) | 10 mg BI 425809 (N=122) | 25 mg BI 425809 (N=123) | Placebo Group (N=120)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg BI 425809 (N=123) | 5 mg BI 425809 (N=122) | 10 mg BI 425809 (N=122) | 25 mg BI 425809 (N=123) | Placebo Group (N=120)
Nausea (Gastrointestinal disorders) | 6 | 1 | 2 | 8 | 2
Nasopharyngitis (Infections and infestations) | 3 | 7 | 3 | 3 | 3
Dizziness (Nervous system disorders) | 4 | 9 | 3 | 6 | 2
Headache (Nervous system disorders) | 6 | 10 | 7 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02788513/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02788513/SAP_001.pdf